CLINICAL TRIAL: NCT03512288
Title: A PHASE 2, RANDOMIZED, DOUBLE-BLIND TRIAL TO EVALUATE THE SAFETY AND IMMUNOGENICITY OF A MULTIVALENT PNEUMOCOCCAL CONJUGATE VACCINE IN HEALTHY INFANTS
Brief Title: Trial to Evaluate the Safety and Immunogenicity of a Multivalent Pneumococcal Vaccine in Healthy Infants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: B7471003
Record Dates: First submitted 2018-04-11; First posted 2018-04-30 (Actual); Results first posted 2021-03-02 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: Pneumococcal Infections
MeSH Terms: conditions — Pneumococcal Infections | interventions — Vaccines, Combined; Pneumococcal Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Multivalent (Experimental): Pneumococcal conjugate vaccines
  Interventions: Biological: Multivalent
- Control (Active Comparator): 13vPnC
  Interventions: Biological: 13vPnC

INTERVENTIONS:
Biological: Multivalent — Pneumococcal conjugate vaccine
  Other Names: Pneumococcal conjugate vaccine
  Arms: Multivalent
Biological: 13vPnC — Pneumococcal conjugate vaccine
  Arms: Control

SUMMARY:
A Phase 2, Randomized, Double-Blind Trial to Evaluate the Safety and Immunogenicity of a Multivalent Pneumococcal Conjugate Vaccine in Healthy Infants

DETAILED DESCRIPTION:
NOTE: Detailed description has not been entered.

ELIGIBILITY:
Inclusion Criteria:

* Male or female infant born at >36 weeks of gestation and aged 2 months (42 to 98 days) at the time of consent (the day of birth is considered day of life 1).
* Healthy infant determined by medical history, physical examination, and clinical judgment to be eligible for the study.

Exclusion Criteria:

* Previous vaccination with licensed or investigational pneumococcal vaccine.
* Prior receipt of diphtheria, tetanus, pertussis, or polio vaccines.
* Previous receipt of >1 dose of hepatitis B vaccine.
* Prior hepatitis B vaccine must have been administered at age <30 days.
* Major known congenital malformation or serious chronic disorder. Receipt of blood/plasma products or immunoglobulins

Ages: 42 Days to 98 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 460 (Actual)
Dates: Start 2018-04-16 (Actual); Primary Completion 2020-02-11 (Actual); Study Completion 2020-02-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (37):
- United States (37):
  - Northwest Arkansas Pediatrics, Fayetteville, Arkansas
  - Premier Health Research Center, LLC, Downey, California
  - St. Joseph Heritage Healthcare, Huntington Beach, California
  - Kaiser Permanente Oakland, Oakland, California
  - Orange County Research Institute, Ontario, California
  - Kaiser Permanente South Sacramento, Sacramento, California
  - Kaiser Permanente San Jose, San Jose, California
  - Kaiser Permanente Santa Clara, Santa Clara, California
  - ACC Pediatric Research, Haughton, Louisiana
  - MedPharmics, LLC, Metairie, Louisiana
  - LSUHSC Shreveport, Shreveport, Louisiana
  - University Health Shreveport, Shreveport, Louisiana
  - Children's Physicians, Creighton University Medical Center, Omaha, Nebraska
  - Child Health Care Associates, East Syracuse, New York
  - Blue Ridge Pediatric and Adolescent Medicine, Inc., Boone, North Carolina
  - Capitol Pediatrics & Adolescent Center PLLC, Raleigh, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Cincinnati Children's Medical Center, Cincinnati, Ohio
  - Pediatric Associates of Mt. Carmel, Inc., Cincinnati, Ohio
  - Ohio Pediatric Research Association, Inc., Dayton, Ohio
  - Senders Pediatrics, South Euclid, Ohio
  - Oklahoma State University - Center for Health Sciences, Tulsa, Oklahoma
  - Allegheny Health and Wellness Pavilion, Erie, Pennsylvania
  - CCP - Kid's Way, Hermitage, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Coastal Pediatric Associates, Charleston, South Carolina
  - Coastal Pediatric Research, Charleston, South Carolina
  - Palmetto Pediatrics, PA, North Charleston, South Carolina
  - University of Texas Medical Branch, Galveston, Texas
  - Tekton Research, Inc., San Antonio, Texas
  - Wee Care Pediatrics, Layton, Utah
  - Wasatch Pediatrics, Cottonwood Office, Murray, Utah
  - Wee Care Pediatrics, Roy, Utah
  - CopperView Medical Center, South Jordan, Utah
  - Wee Care Pediatrics, Syracuse, Utah
  - Pediatric Associates of Charlottesville, PLC, Charlottesville, Virginia
  - Pediatric Research of Charlottesville, LLC, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Senders S, Klein NP, Lamberth E, Thompson A, Drozd J, Trammel J, Peng Y, Giardina PC, Jansen KU, Gruber WC, Scott DA, Watson W. Safety and Immunogenicity of a 20-valent Pneumococcal Conjugate Vaccine in Healthy Infants in the United States. Pediatr Infect Dis J. 2021 Oct 1;40(10):944-951. doi: 10.1097/INF.0000000000003277. PMID 34525007
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7471003

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 16 April 2018 to 11 February 2020 in the United States.
Pre-assignment Details: A total of 460 participants of age greater than or equal to (>=) 42 to less than or equal to (<=) 98 days at baseline, were enrolled into the study. Out of these 460 participants, 458 participants received study treatment.
Groups:
- 20vPnC: Participants were randomized to receive a single 0.5 milliliter (mL) intramuscular injection of 20-valent pneumococcal conjugate vaccine (20vPnC) at 2, 4, 6, and 12 months of age (Dose/Vaccination 1, 2, 3, and 4 respectively).
- 13vPnC: Participants were randomized to receive a single 0.5 mL intramuscular injection of 13-valent pneumococcal conjugate vaccine (13vPnC) at 2, 4, 6, and 12 months of age (Dose/Vaccination 1, 2, 3, and 4, respectively).
Period: Overall Study
Arm/Group | 20vPnC | 13vPnC
Started | 232 | 228
Vaccination 1 | 231 | 227
Vaccination 2 | 222 | 213
Vaccination 3 | 210 | 206
Vaccination 4 | 197 | 194
Completed | 191 | 185
Not Completed | 41 | 43
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 12 | 15
Not completed — Physician Decision | 0 | 2
Not completed — Protocol Violation | 6 | 4
Not completed — Medication error without associated adverse event | 1 | 0
Not completed — No longer met eligibility criteria | 5 | 2
Not completed — Withdrawal by parent/guardian | 14 | 18
Not completed — Other | 1 | 1
Not completed — Randomized but not treated | 1 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- 20vPnC: Participants were randomized to receive a single 0.5 mL intramuscular injection of 20vPnC at 2, 4, 6, and 12 months of age (Dose/Vaccination 1, 2, 3, and 4 respectively).
- 13vPnC: Participants were randomized to receive a single 0.5 mL intramuscular injection of 13vPnC at 2, 4, 6, and 12 months of age (Dose/Vaccination 1, 2, 3, and 4, respectively).
- Total: Total of all reporting groups
Arm/Group | 20vPnC | 13vPnC | Total
Number analyzed (Participants) | 232 | 228 | 460
Age, Continuous [Mean (Standard Deviation); unit: days] | 64.5 (8.07) | 64.5 (6.68) | 64.5 (7.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 112 | 115 | 227
  Male | 120 | 113 | 233
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 41 | 40 | 81
  Not Hispanic or Latino | 191 | 188 | 379
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 3 | 7
  Asian | 9 | 5 | 14
  Native Hawaiian or Other Pacific Islander | 1 | 3 | 4
  Black or African American | 35 | 29 | 64
  White | 161 | 171 | 332
  More than one race | 22 | 15 | 37
  Unknown or Not Reported | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Local Reactions Within 7 Days After Vaccination 1
Description: Local reactions were recorded using an electronic diary. Local reactions included redness, swelling and pain at the injection site. Redness and swelling were measured and recorded in measuring device units. 1 measuring device unit =0.5 centimeter (cm). Redness and swelling were graded as mild (0.5 to 2.0 centimeter [cm]), moderate (greater than [>] 2.0 to 7.0 cm) and severe (>7.0 cm). Pain at injection site was graded as mild (hurt if gently touched example, whimpered, winced, protested, or withdrew), moderate (hurt if gently touched, with crying), and severe (caused limitation of limb movement).
Time Frame: Within 7 days after Vaccination 1
Population: Dose 1 to Dose 3 safety population included participants who received Dose 1 and had safety follow up between Dose 1 and the blood draw visit 1 month after Dose 3. Here, "Overall Number of Participants Analyzed" =participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 20vPnC | 13vPnC
Number analyzed (Participants) | 229 | 224
percentage of participants
  Redness: Any | 24.9 [19.4 to 31.0] | 25.4 [19.9 to 31.7]
  Redness: Mild | 22.3 [17.1 to 28.2] | 23.7 [18.3 to 29.8]
  Redness: Moderate | 2.6 [1.0 to 5.6] | 1.8 [0.5 to 4.5]
  Redness: Severe | 0 [0.0 to 1.6] | 0 [0.0 to 1.6]
  Swelling: Any | 12.7 [8.6 to 17.7] | 14.3 [10.0 to 19.6]
  Swelling: Mild | 10.0 [6.5 to 14.7] | 12.9 [8.8 to 18.1]
  Swelling: Moderate | 2.2 [0.7 to 5.0] | 1.3 [0.3 to 3.9]
  Swelling: Severe | 0.4 [0.0 to 2.4] | 0 [0.0 to 1.6]
  Pain at the injection site: Any | 51.1 [44.4 to 57.7] | 53.6 [46.8 to 60.2]
  Pain at the injection site: Mild | 32.3 [26.3 to 38.8] | 35.7 [29.4 to 42.4]
  Pain at the injection site: Moderate | 18.3 [13.5 to 24.0] | 17.9 [13.1 to 23.5]
  Pain at the injection site: Severe | 0.4 [0.0 to 2.4] | 0 [0.0 to 1.6]

2. Primary Outcome: Percentage of Participants With Local Reactions Within 7 Days After Vaccination 2
Description: Local reactions were recorded using an electronic diary. Local reactions included redness, swelling and pain at the injection site. Redness and swelling were measured and recorded in measuring device units. 1 measuring device unit =0.5 cm. Redness and swelling were graded as mild (0.5 to 2.0 cm), moderate (>2.0 to 7.0 cm) and severe (>7.0 cm). Pain at injection site was graded as mild (hurt if gently touched example, whimpered, winced, protested, or withdrew), moderate (hurt if gently touched, with crying), and severe (caused limitation of limb movement).
Time Frame: Within 7 days after Vaccination 2
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 20vPnC | 13vPnC
Number analyzed (Participants) | 215 | 204
percentage of participants
  Redness: Any | 24.7 [19.0 to 31.0] | 28.4 [22.4 to 35.2]
  Redness: Mild | 21.9 [16.5 to 28.0] | 24.0 [18.3 to 30.5]
  Redness: Moderate | 2.8 [1.0 to 6.0] | 4.4 [2.0 to 8.20]
  Redness: Severe | 0 [0.0 to 1.7] | 0 [0.0 to 1.8]
  Swelling: Any | 16.3 [11.6 to 21.9] | 18.6 [13.5 to 24.7]
  Swelling: Mild | 12.6 [8.4 to 17.7] | 13.2 [8.9 to 18.7]
  Swelling: Moderate | 3.7 [1.6 to 7.2] | 5.4 [2.7 to 9.4]
  Swelling: Severe | 0 [0.0 to 1.7] | 0 [0.0 to 1.8]
  Pain at the injection site: Any | 42.8 [36.1 to 49.7] | 48.5 [41.5 to 55.6]
  Pain at the injection site: Mild | 26.0 [20.3 to 32.5] | 28.9 [22.8 to 35.7]
  Pain at the injection site: Moderate | 15.8 [11.2 to 21.4] | 19.6 [14.4 to 25.7]
  Pain at the injection site: Severe | 0.9 [0.1 to 3.3] | 0 [0.0 to 1.8]

3. Primary Outcome: Percentage of Participants With Local Reactions Within 7 Days After Vaccination 3
Description: as for outcome 2
Time Frame: Within 7 days after Vaccination 3
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 20vPnC | 13vPnC
Number analyzed (Participants) | 201 | 204
percentage of participants
  Redness: Any | 26.9 [20.9 to 33.6] | 26.5 [20.6 to 33.1]
  Redness: Mild | 26.4 [20.4 to 33.0] | 23.0 [17.4 to 29.4]
  Redness: Moderate | 0.5 [0.0 to 2.7] | 3.4 [1.4 to 6.9]
  Redness: Severe | 0 [0.0 to 1.8] | 0 [0.0 to 1.8]
  Swelling: Any | 17.9 [12.9 to 23.9] | 19.6 [14.4 to 25.7]
  Swelling: Mild | 16.9 [12.0 to 22.8] | 15.7 [11.0 to 21.4]
  Swelling: Moderate | 1.0 [0.1 to 3.5] | 3.4 [1.4 to 6.9]
  Swelling: Severe | 0 [0.0 to 1.8] | 0.5 [0.0 to 2.7]
  Pain at the injection site: Any | 44.3 [37.3 to 51.4] | 40.7 [33.9 to 47.8]
  Pain at the injection site: Mild | 28.9 [22.7 to 35.6] | 27.9 [21.9 to 34.6]
  Pain at the injection site: Moderate | 14.9 [10.3 to 20.6] | 12.7 [8.5 to 18.1]
  Pain at the injection site: Severe | 0.5 [0.0 to 2.7] | 0 [0.0 to 1.8]

4. Primary Outcome: Percentage of Participants With Local Reactions Within 7 Days After Vaccination 4
Description: as for outcome 2
Time Frame: Within 7 days after Vaccination 4
Population: Dose 4 safety population included participants who received Dose 4 and had safety follow up between Dose 4 and 6 months after Dose 4. Here, "Overall Number of Participants Analyzed" =participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 20vPnC | 13vPnC
Number analyzed (Participants) | 186 | 185
percentage of participants
  Redness: Any | 25.8 [19.7 to 32.7] | 30.3 [23.7 to 37.4]
  Redness: Mild | 24.2 [18.2 to 31.0] | 25.4 [19.3 to 32.3]
  Redness: Moderate | 1.6 [0.3 to 4.6] | 4.9 [2.2 to 9.0]
  Redness: Severe | 0 [0.0 to 2.0] | 0 [0.0 to 2.0]
  Swelling: Any | 17.2 [12.1 to 23.4] | 14.1 [9.4 to 19.9]
  Swelling: Mild | 15.1 [10.2 to 21.0] | 12.4 [8.0 to 18.1]
  Swelling: Moderate | 2.2 [0.6 to 5.4] | 1.6 [0.3 to 4.7]
  Swelling: Severe | 0 [0.0 to 2.0] | 0 [0.0 to 2.0]
  Pain at the injection site: Any | 35.5 [28.6 to 42.8] | 35.7 [28.8 to 43.0]
  Pain at the injection site: Mild | 26.9 [20.7 to 33.9] | 28.6 [22.3 to 35.7]
  Pain at the injection site: Moderate | 8.6 [5.0 to 13.6] | 7.0 [3.8 to 11.7]
  Pain at the injection site: Severe | 0 [0.0 to 2.0] | 0 [0.0 to 2.0]

5. Primary Outcome: Percentage of Participants With Systemic Events Within 7 Days After Vaccination 1
Description: Systemic events included fever, decreased appetite, drowsiness, irritability and were recorded by using an electronic diary. Fever was defined as greater than or equal to (>=) 38.0 degree Celsius (C) and categorized to >=38.0 to 38.4 degree C, >38.4 to 38.9 degree C, >38.9 to 40.0 degree C and >40.0 degree C. Decreased appetite was graded as mild (decreased interest in eating), moderate (decreased oral intake) and severe (refusal to feed). Drowsiness was graded as mild (increased or prolonged sleeping bouts), moderate (slightly subdued, interfered with daily activity) and severe (disabled, not interested in usual daily activity). Irritability was graded as mild (easily consolable), moderate (required increased attention) and severe (inconsolable; crying could not be comforted).
Time Frame: Within 7 days after Vaccination 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 20vPnC | 13vPnC
Number analyzed (Participants) | 229 | 224
percentage of participants
  Fever: >=38.0 degree C | 14.4 [10.1 to 19.6] | 9.8 [6.3 to 14.5]
  Fever: >=38.0 degree C to 38.4 degree C | 10.0 [6.5 to 14.7] | 6.3 [3.5 to 10.3]
  Fever: >38.4 degree C to 38.9 degree C | 3.9 [1.8 to 7.3] | 2.2 [0.7 to 5.1]
  Fever: >38.9 degree C to 40.0 degree C | 0.4 [0.0 to 2.4] | 1.3 [0.3 to 3.9]
  Fever: >40.0 degree C | 0 [0.0 to 1.6] | 0 [0.0 to 1.6]
  Decreased appetite: Any | 25.3 [19.8 to 31.5] | 30.4 [24.4 to 36.8]
  Decreased appetite: Mild | 16.2 [11.6 to 21.6] | 19.2 [14.3 to 25.0]
  Decreased appetite: Moderate | 9.2 [5.8 to 13.7] | 10.7 [7.0 to 15.5]
  Decreased appetite: Severe | 0 [0.0 to 1.6] | 0.4 [0.0 to 2.5]
  Drowsiness: Any | 68.1 [61.7 to 74.1] | 71.0 [64.6 to 76.8]
  Drowsiness: Mild | 51.1 [44.4 to 57.7] | 54.9 [48.1 to 61.5]
  Drowsiness: Moderate | 16.6 [12.0 to 22.1] | 14.3 [10.0 to 19.6]
  Drowsiness: Severe | 0.4 [0.0 to 2.4] | 1.8 [0.5 to 4.5]
  Irritability: Any | 79.5 [73.7 to 84.5] | 77.7 [71.7 to 83.0]
  Irritability: Mild | 23.6 [18.2 to 29.6] | 25.9 [20.3 to 32.1]
  Irritability: Moderate | 50.7 [44.0 to 57.3] | 47.3 [40.6 to 54.1]
  Irritability: Severe | 5.2 [2.7 to 9.0] | 4.5 [2.2 to 8.1]

6. Primary Outcome: Percentage of Participants With Systemic Events Within 7 Days After Vaccination 2
Description: Systemic events included fever, decreased appetite, drowsiness, irritability and were recorded by using an electronic diary. Fever was defined as >= 38.0 degree Celsius (C) and categorized to >=38.0 to 38.4 degree C, >38.4 to 38.9 degree C, >38.9 to 40.0 degree C and >40.0 degree C. Decreased appetite was graded as mild (decreased interest in eating), moderate (decreased oral intake) and severe (refusal to feed). Drowsiness was graded as mild (increased or prolonged sleeping bouts), moderate (slightly subdued, interfered with daily activity) and severe (disabled, not interested in usual daily activity). Irritability was graded as mild (easily consolable), moderate (required increased attention) and severe (inconsolable; crying could not be comforted).
Time Frame: Within 7 days after Vaccination 2
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 20vPnC | 13vPnC
Number analyzed (Participants) | 215 | 204
percentage of participants
  Fever: >=38.0 degree C | 17.2 [12.4 to 22.9] | 23.0 [17.4 to 29.4]
  Fever: >=38.0 degree C to 38.4 degree C | 10.2 [6.5 to 15.1] | 12.7 [8.5 to 18.1]
  Fever: >38.4 degree C to 38.9 degree C | 4.2 [1.9 to 7.8] | 7.8 [4.5 to 12.4]
  Fever: >38.9 degree C to 40.0 degree C | 2.8 [1.0 to 6.0] | 2.5 [0.8 to 5.6]
  Fever: >40.0 degree C | 0 [0.0 to 1.7] | 0 [0.0 to 1.8]
  Decreased appetite: Any | 23.3 [17.8 to 29.5] | 27.0 [21.0 to 33.6]
  Decreased appetite: Mild | 14.4 [10.0 to 19.8] | 14.7 [10.1 to 20.3]
  Decreased appetite: Moderate | 7.9 [4.7 to 12.4] | 11.8 [7.7 to 17.0]
  Decreased appetite: Severe | 0.9 [0.1 to 3.3] | 0.5 [0.0 to 2.7]
  Drowsiness: Any | 57.2 [50.3 to 63.9] | 56.4 [49.3 to 63.3]
  Drowsiness: Mild | 37.2 [30.7 to 44.0] | 37.7 [31.1 to 44.8]
  Drowsiness: Moderate | 17.7 [12.8 to 23.4] | 16.7 [11.8 to 22.5]
  Drowsiness: Severe | 2.3 [0.8 to 5.3] | 2.0 [0.5 to 4.9]
  Irritability: Any | 71.2 [64.6 to 77.1] | 79.9 [73.7 to 85.2]
  Irritability: Mild | 20.0 [14.9 to 26.0] | 22.5 [17.0 to 28.9]
  Irritability: Moderate | 48.8 [42.0 to 55.7] | 52.5 [45.4 to 59.5]
  Irritability: Severe | 2.3 [0.8 to 5.3] | 4.9 [2.4 to 8.8]

7. Primary Outcome: Percentage of Participants With Systemic Events Within 7 Days After Vaccination 3
Description: as for outcome 6
Time Frame: Within 7 days after Vaccination 3
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 20vPnC | 13vPnC
Number analyzed (Participants) | 201 | 204
percentage of participants
  Fever: >=38.0 degree C | 17.9 [12.9 to 23.9] | 18.1 [13.1 to 24.1]
  Fever: >=38.0 degree C to 38.4 degree C | 10.0 [6.2 to 14.9] | 9.8 [6.1 to 14.7]
  Fever: >38.4 degree C to 38.9 degree C | 4.5 [2.1 to 8.3] | 4.9 [2.4 to 8.8]
  Fever: >38.9 degree C to 40.0 degree C | 3.5 [1.4 to 7.0] | 3.4 [1.4 to 6.9]
  Fever: >40.0 degree C | 0 [0.0 to 1.8] | 0 [0.0 to 1.8]
  Decreased appetite: Any | 30.8 [24.5 to 37.7] | 33.3 [26.9 to 40.3]
  Decreased appetite: Mild | 20.9 [15.5 to 27.2] | 19.1 [14.0 to 25.2]
  Decreased appetite: Moderate | 9.5 [5.8 to 14.4] | 13.7 [9.3 to 19.2]
  Decreased appetite: Severe | 0.5 [0.0 to 2.7] | 0.5 [0.0 to 2.7]
  Drowsiness: Any | 41.3 [34.4 to 48.4] | 45.6 [38.6 to 52.7]
  Drowsiness: Mild | 28.9 [22.7 to 35.6] | 29.9 [23.7 to 36.7]
  Drowsiness: Moderate | 11.4 [7.4 to 16.7] | 15.7 [11.0 to 21.4]
  Drowsiness: Severe | 1.0 [0.1 to 3.5] | 0 [0.0 to 1.8]
  Irritability: Any | 72.6 [65.9 to 78.7] | 69.6 [62.8 to 75.8]
  Irritability: Mild | 28.9 [22.7 to 35.6] | 27.5 [21.5 to 34.1]
  Irritability: Moderate | 40.8 [33.9 to 47.9] | 37.7 [31.1 to 44.8]
  Irritability: Severe | 3.0 [1.1 to 6.4] | 4.4 [2.0 to 8.2]

8. Primary Outcome: Percentage of Participants With Systemic Events Within 7 Days After Vaccination 4
Description: as for outcome 6
Time Frame: Within 7 days after Vaccination 4
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 20vPnC | 13vPnC
Number analyzed (Participants) | 186 | 185
percentage of participants
  Fever: >=38.0 degree C | 12.4 [8.0 to 18.0] | 14.6 [9.8 to 20.5]
  Fever: >=38.0 degree C to 38.4 degree C | 5.9 [3.0 to 10.3] | 4.3 [1.9 to 8.3]
  Fever: >38.4 degree C to 38.9 degree C | 3.2 [1.2 to 6.9] | 7.0 [3.8 to 11.7]
  Fever: >38.9 degree C to 40.0 degree C | 3.2 [1.2 to 6.9] | 3.2 [1.2 to 6.9]
  Fever: >40.0 degree C | 0 [0.0 to 2.0] | 0 [0.0 to 2.0]
  Decreased appetite: Any | 23.7 [17.7 to 30.4] | 29.2 [22.8 to 36.3]
  Decreased appetite: Mild | 13.4 [8.9 to 19.2] | 15.7 [10.8 to 21.7]
  Decreased appetite: Moderate | 10.2 [6.3 to 15.5] | 13.5 [8.9 to 19.3]
  Decreased appetite: Severe | 0 [0.0 to 2.0] | 0 [0.0 to 2.0]
  Drowsiness: Any | 32.8 [26.1 to 40.0] | 37.3 [30.3 to 44.7]
  Drowsiness: Mild | 26.9 [20.7 to 33.9] | 25.4 [19.3 to 32.3]
  Drowsiness: Moderate | 4.8 [2.2 to 9.0] | 11.9 [7.6 to 17.4]
  Drowsiness: Severe | 1.1 [0.1 to 3.8] | 0 [0.0 to 2.0]
  Irritability: Any | 62.4 [55.0 to 69.3] | 62.7 [55.3 to 69.7]
  Irritability: Mild | 23.7 [17.7 to 30.4] | 19.5 [14.0 to 25.9]
  Irritability: Moderate | 36.0 [29.1 to 43.4] | 40.0 [32.9 to 47.4]
  Irritability: Severe | 2.7 [0.9 to 6.2] | 3.2 [1.2 to 6.9]

9. Primary Outcome: Percentage of Participants With Adverse Events (AEs) From Vaccination 1 to 1 Month After Vaccination 3
Description: An AE was any untoward medical occurrence in study participants who received study vaccine without regard to possibility of causal relationship.
Time Frame: From Vaccination 1 to 1 month after Vaccination 3 (up to 5 months)
Population: Dose 1 to Dose 3 safety population included participants who received Dose 1 and had safety follow up between Dose 1 and the blood draw visit 1 month after Dose 3.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 20vPnC | 13vPnC
Number analyzed (Participants) | 231 | 227
percentage of participants | 61.0 [54.4 to 67.4] | 56.4 [49.7 to 62.9]

10. Primary Outcome: Percentage of Participants With Adverse Events (AEs) From Vaccination 4 to 1 Month After Vaccination 4
Description: An AE was any untoward medical occurrence in study participant who received study vaccine without regard to possibility of causal relationship.
Time Frame: From Vaccination 4 to 1 month after Vaccination 4
Population: Dose 4 safety population included participants who received Dose 4 and had safety follow up between Dose 4 and 6 months after Dose 4.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 20vPnC | 13vPnC
Number analyzed (Participants) | 197 | 194
percentage of participants | 18.3 [13.1 to 24.4] | 25.3 [19.3 to 32.0]

11. Primary Outcome: Percentage of Participants With Serious Adverse Events (SAEs) From Vaccination 1 to 6 Months Following Vaccination 4
Description: An SAE is any untoward medical occurrence at any dose that results in death; is life-threatening (immediate risk of death); requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity (substantial disruption of the ability to conduct normal life functions); results in congenital anomaly/birth defect.
Time Frame: From Vaccination 1 to 6 months after Vaccination 4 (up to 16 months)
Population: Overall safety analysis set included all participants who received at least 1 dose of study vaccine (20vPnC or 13vPnC) and had safety follow up in the study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 20vPnC | 13vPnC
Number analyzed (Participants) | 231 | 227
percentage of participants | 5.2 [2.7 to 8.9] | 2.2 [0.7 to 5.1]

12. Primary Outcome: Percentage of Participants With Newly Diagnosed Chronic Medical Conditions (NDCMCs) From Vaccination 1 to 6 Months Following Vaccination 4
Description: An NDCMC is defined as a disease or medical condition, not previously identified, that is expected to be persistent or is otherwise long-lasting in its effects.
Time Frame: From Vaccination 1 to 6 months after Vaccination 4 (duration of 16 months)
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 20vPnC | 13vPnC
Number analyzed (Participants) | 231 | 227
percentage of participants | 5.2 [2.7 to 8.9] | 3.5 [1.5 to 6.8]

13. Secondary Outcome: Percentage of Participants Who Achieved Pre-specified Level of Pneumococcal IgG Concentrations Within 1 Month After Vaccination 3
Description: Pre-specified levels of serotypes were as follows: for serotype 1, 3, 4, 6A, 7F, 9V, 14, 18C, 19F, 23F, 8, 10A, 11A, 12F, 15B, 22F, 33F: >=0.35 microgram per milliliter, for serotype 5: >=0.23 microgram per milliliter, for serotype 6B: >=0.10 microgram per milliliter and for serotype 19A: >=0.12 microgram per milliliter.
Time Frame: 1 month after Vaccination 3
Population: Dose 3 evaluable immunogenicity population: included all eligible participants, who were randomly assigned to receive the vaccine, aged 42-98 days on the day of first vaccination, received 3 doses of assigned vaccine, had valid determinate IgG concentration for at least 1 serotype from 1 month after Dose 3 visit, had blood collection within 27-56 days, inclusive, after Dose 3, had not received prohibited vaccines before blood draw at 1 month after Dose 3, and had no major protocol deviations.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 20vPnC | 13vPnC
Number analyzed (Participants) | 189 | 187
percentage of participants
  Serotype 1 | 87.8 [82.3 to 92.1] | 87.7 [82.1 to 92.0]
  Serotype 3 | 65.1 [57.8 to 71.9] | 75.4 [68.6 to 81.4]
  Serotype 4 | 87.8 [82.3 to 92.1] | 91.4 [86.5 to 95.0]
  Serotype 5 | 87.8 [82.3 to 92.1] | 89.8 [84.6 to 93.8]
  Serotype 6A | 93.7 [89.2 to 96.7] | 92.5 [87.8 to 95.8]
  Serotype 6B | 86.8 [81.1 to 91.3] | 90.4 [85.2 to 94.2]
  Serotype 7F | 98.9 [96.2 to 99.9] | 97.9 [94.6 to 99.4]
  Serotype 9V | 89.4 [84.1 to 93.4] | 89.3 [84.0 to 93.3]
  Serotype 14 | 94.2 [89.8 to 97.1] | 95.7 [91.7 to 98.1]
  Serotype 18C | 92.6 [87.9 to 95.9] | 95.2 [91.1 to 97.8]
  Serotype 19A | 98.4 [95.4 to 99.7] | 97.9 [94.6 to 99.4]
  Serotype 19F | 98.4 [95.4 to 99.7] | 96.8 [93.1 to 98.8]
  Serotype 23F | 79.9 [73.5 to 85.4] | 81.8 [75.5 to 87.1]
  Serotype 8 | 99.5 [97.1 to 100.0] | 3.7 [1.5 to 7.6]
  Serotype 10A | 87.8 [82.3 to 92.1] | 1.1 [0.1 to 3.8]
  Serotype 11A | 97.4 [93.9 to 99.1] | 1.6 [0.3 to 4.6]
  Serotype 12F | 82.5 [76.4 to 87.7] | 0.5 [0.0 to 2.9]
  Serotype 15B | 98.9 [96.2 to 99.9] | 4.3 [1.9 to 8.3]
  Serotype 22F | 98.9 [96.2 to 99.9] | 1.1 [0.1 to 3.8]
  Serotype 33F | 92.1 [87.2 to 95.5] | 1.6 [0.3 to 4.6]

14. Secondary Outcome: Pneumococcal Serotype-specific Immunoglobulin G (IgG) Geometric Mean Concentrations (GMCs) at 1 Month After Vaccination 3
Description: IgG GMCs were determined for each of the 20 pneumococcal serotypes 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, 23F, 8, 10A, 11A, 12F, 15B, 22F and 33F.
Time Frame: 1 month after Vaccination 3
Population: as for outcome 13
Measure: Geometric Mean (95% Confidence Interval); unit: microgram per milliliter
Arm/Group | 20vPnC | 13vPnC
Number analyzed (Participants) | 189 | 187
microgram per milliliter
  Serotype 1 | 0.92 [0.81 to 1.05] | 1.16 [1.00 to 1.33]
  Serotype 3 | 0.43 [0.38 to 0.48] | 0.56 [0.49 to 0.64]
  Serotype 4 | 1.36 [1.16 to 1.61] | 1.64 [1.39 to 1.93]
  Serotype 5 | 0.93 [0.79 to 1.11] | 1.13 [0.96 to 1.34]
  Serotype 6A | 2.28 [1.94 to 2.67] | 2.57 [2.16 to 3.05]
  Serotype 6B | 0.63 [0.49 to 0.80] | 0.99 [0.77 to 1.27]
  Serotype 7F | 2.15 [1.92 to 2.40] | 2.59 [2.28 to 2.93]
  Serotype 9V | 1.22 [1.05 to 1.42] | 1.45 [1.24 to 1.70]
  Serotype 14 | 3.15 [2.69 to 3.70] | 3.60 [3.07 to 4.21]
  Serotype 18C | 1.59 [1.37 to 1.84] | 2.05 [1.76 to 2.38]
  Serotype 19A | 0.85 [0.74 to 0.96] | 1.02 [0.89 to 1.17]
  Serotype 19F | 1.98 [1.76 to 2.22] | 2.28 [1.99 to 2.61]
  Serotype 23F | 0.94 [0.78 to 1.14] | 1.26 [1.03 to 1.55]
  Serotype 8 | 2.09 [1.90 to 2.30] | 0.04 [0.03 to 0.04]
  Serotype 10A | 1.67 [1.35 to 2.08] | 0.03 [0.03 to 0.03]
  Serotype 11A | 1.94 [1.70 to 2.21] | 0.01 [0.01 to 0.01]
  Serotype 12F | 0.86 [0.72 to 1.01] | 0.02 [0.02 to 0.02]
  Serotype 15B | 5.86 [5.11 to 6.72] | 0.04 [0.04 to 0.05]
  Serotype 22F | 4.62 [3.99 to 5.35] | 0.01 [0.01 to 0.01]
  Serotype 33F | 2.21 [1.87 to 2.61] | 0.05 [0.04 to 0.05]

15. Secondary Outcome: Pneumococcal Serotype-specific IgG GMCs at 1 Month After Vaccination 4
Description: as for outcome 14
Time Frame: 1 Month after Vaccination 4
Population: Dose 4 evaluable immunogenicity population: eligible participants, randomly assigned to receive vaccine, aged 42-98 days on day of first vaccination, received all 4 doses of assigned vaccine, with Dose 4 received in defined window (365-386 days of age), had valid determinate IgG concentration for at least 1 serotype 1 month post dose 4,had blood collection within 27-56 days post Dose 4,had not received prohibited vaccines before blood draw at 1 month post Dose 4,had no major protocol deviations.
Measure: Geometric Mean (95% Confidence Interval); unit: microgram per milliliter
Arm/Group | 20vPnC | 13vPnC
Number analyzed (Participants) | 168 | 166
microgram per milliliter
  Serotype 1 | 2.65 [2.33 to 3.02] | 3.63 [3.20 to 4.11]
  Serotype 3 | 1.15 [0.97 to 1.35] | 1.49 [1.28 to 1.74]
  Serotype 4 | 7.16 [6.22 to 8.24] | 9.45 [8.16 to 10.95]
  Serotype 5 | 3.41 [2.95 to 3.93] | 4.95 [4.29 to 5.71]
  Serotype 6A | 13.77 [12.16 to 15.59] | 18.83 [16.39 to 21.63]
  Serotype 6B | 6.37 [5.42 to 7.50] | 9.73 [8.13 to 11.65]
  Serotype 7F | 6.14 [5.51 to 6.83] | 9.32 [8.26 to 10.52]
  Serotype 9V | 5.52 [4.82 to 6.31] | 7.78 [6.77 to 8.95]
  Serotype 14 | 8.61 [7.32 to 10.12] | 11.04 [9.44 to 12.90]
  Serotype 18C | 5.58 [4.89 to 6.36] | 8.46 [7.25 to 9.88]
  Serotype 19A | 5.71 [4.91 to 6.64] | 7.05 [6.04 to 8.24]
  Serotype 19F | 7.79 [6.73 to 9.01] | 9.30 [7.99 to 10.83]
  Serotype 23F | 6.06 [5.16 to 7.12] | 9.81 [8.10 to 11.88]
  Serotype 8 | 3.12 [2.78 to 3.49] | 0.05 [0.04 to 0.06]
  Serotype 10A | 9.93 [8.58 to 11.50] | 0.03 [0.03 to 0.04]
  Serotype 11A | 5.70 [4.96 to 6.54] | 0.01 [0.01 to 0.02]
  Serotype 12F | 1.92 [1.68 to 2.20] | 0.02 [0.02 to 0.03]
  Serotype 15B | 18.45 [16.43 to 20.72] | 0.04 [0.04 to 0.05]
  Serotype 22F | 14.68 [12.62 to 17.08] | 0.01 [0.01 to 0.01]
  Serotype 33F | 4.70 [4.20 to 5.27] | 0.05 [0.04 to 0.05]

ADVERSE EVENTS:
Time Frame: Local reactions and Systemic events: within 7 days after each vaccination (systematic assessment), Non serious AEs: Vaccination 1 to 1 month after Vaccination 3 (up to 5 months) and Vaccination 4 to 1 month after Vaccination 4, SAEs: up to 16 months after Vaccination 1
Description: Same event may appear as AE and SAE, what is presented are distinct events. Event may be categorized as serious in 1 participant and as non-serious in another participant or 1 participant may have experienced both serious and non-serious event during study. Overall safety analysis set was analyzed.
Arm/Group | 20vPnC | 13vPnC
All-Cause Mortality (participants affected / at risk) | 0/231 | 0/227
Serious Adverse Events (participants affected / at risk) | 12/231 | 5/227
Other Adverse Events (participants affected / at risk) | 225/231 | 224/227
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 20vPnC (N=231) | 13vPnC (N=227)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Bronchiolitis (Infections and infestations) | 1 | 0
Bronchitis viral (Infections and infestations) | 1 | 0
Croup infectious (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 1
Meningitis viral (Infections and infestations) | 1 | 0
Parainfluenzae virus infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 1 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0
Seizure like phenomena (Nervous system disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oliguria (Renal and urinary disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 20vPnC (N=231) | 13vPnC (N=227)
Plagiocephaly (Congenital, familial and genetic disorders) | 2 | 4
Ear pain (Ear and labyrinth disorders) | 3 | 2
Constipation (Gastrointestinal disorders) | 10 | 6
Diarrhoea (Gastrointestinal disorders) | 10 | 10
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 6 | 10
Haematochezia (Gastrointestinal disorders) | 0 | 3
Teething (Gastrointestinal disorders) | 10 | 16
Vomiting (Gastrointestinal disorders) | 8 | 9
Injection site erythema (REDNESS) (General disorders) | 112 | 120
Injection site pain (PAIN) (General disorders) | 163 | 167
Injection site swelling (SWELLING) (General disorders) | 76 | 81
Pyrexia (General disorders) | 12 | 10
Food allergy (Immune system disorders) | 0 | 3
Bronchiolitis (Infections and infestations) | 11 | 11
Candida infection (Infections and infestations) | 4 | 5
Candida nappy rash (Infections and infestations) | 0 | 5
Cellulitis (Infections and infestations) | 3 | 1
Conjunctivitis (Infections and infestations) | 12 | 11
Conjunctivitis bacterial (Infections and infestations) | 3 | 0
Ear infection (Infections and infestations) | 2 | 4
Gastroenteritis (Infections and infestations) | 2 | 8
Gastroenteritis viral (Infections and infestations) | 6 | 1
Hand-foot-and-mouth disease (Infections and infestations) | 1 | 3
Nasopharyngitis (Infections and infestations) | 15 | 16
Oral candidiasis (Infections and infestations) | 3 | 3
Otitis media (Infections and infestations) | 25 | 21
Otitis media acute (Infections and infestations) | 8 | 15
Pneumonia (Infections and infestations) | 3 | 0
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 2 | 3
Respiratory tract infection viral (Infections and infestations) | 6 | 4
Skin candida (Infections and infestations) | 0 | 5
Upper respiratory tract infection (Infections and infestations) | 40 | 44
Viral infection (Infections and infestations) | 10 | 10
Viral upper respiratory tract infection (Infections and infestations) | 15 | 11
Fall (Injury, poisoning and procedural complications) | 6 | 2
Decreased appetite (DECREASED APPETITE) (Metabolism and nutrition disorders) | 134 | 136
Failure to thrive (Metabolism and nutrition disorders) | 2 | 3
Feeding disorder (Metabolism and nutrition disorders) | 2 | 3
Acquired plagiocephaly (Musculoskeletal and connective tissue disorders) | 1 | 4
Torticollis (Musculoskeletal and connective tissue disorders) | 3 | 2
Agitation neonatal (Nervous system disorders) | 2 | 4
Hypersomnia (INCREASED SLEEP) (Nervous system disorders) | 188 | 189
Irritability (IRRITABILITY) (Psychiatric disorders) | 214 | 206
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 8
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 12 | 7
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 6 | 5
Dermatitis contact (Skin and subcutaneous tissue disorders) | 3 | 0
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 11 | 8
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 3
Eczema (Skin and subcutaneous tissue disorders) | 5 | 3
Eczema infantile (Skin and subcutaneous tissue disorders) | 1 | 3
Rash (Skin and subcutaneous tissue disorders) | 5 | 5
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 4
Croup infectious (Infections and infestations) | 4 | 3
Pyrexia (FEVER) (General disorders) | 90 | 90

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-04-12): https://cdn.clinicaltrials.gov/large-docs/88/NCT03512288/SAP_000.pdf
  • Study Protocol (2020-02-11): https://cdn.clinicaltrials.gov/large-docs/88/NCT03512288/Prot_001.pdf